CLINICAL TRIAL: NCT02584543
Title: Safety and Immunogenicity Study of the Recombinant Hepatitis E Vaccine(Escherichia Coli) Coadministration With Recombinant Hepatitis B Vaccine
Brief Title: A Phase Ⅳ Clinical Trial of the Recombinant Hepatitis E Vaccine (Escherichia Coli)(Coadministration With Recombinant Hepatitis B Vaccine)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-HE-007
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis E; Hepatitis B
MeSH Terms: conditions — Hepatitis E; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HEV vaccine and HBV vaccine Co-administration group (Experimental)
  Interventions: Biological: HEV vaccine; Biological: HBV vaccine
- HEV vaccine control group (Active Comparator)
  Interventions: Biological: HEV vaccine
- HBV vaccine control group (Active Comparator)
  Interventions: Biological: HBV vaccine

INTERVENTIONS:
Biological: HEV vaccine
  Arms: HEV vaccine and HBV vaccine Co-administration group; HEV vaccine control group
Biological: HBV vaccine
  Arms: HBV vaccine control group; HEV vaccine and HBV vaccine Co-administration group

SUMMARY:
This is a open label, randomized phase VI study, to assess the safety and immunogenicity of co-administration of Hepatitis E vaccine with Hepatitis B vaccine. The concomitant group (n =300) received Hepatitis B vaccine concomitantly with Hepatitis E vaccine at day 1 and months 1 and 6; The nonconcomitant group (n =150) received Hepatitis E vaccine at at day 1 and months 1 and 6. Another nonconcomitant group (n=150) received Hepatitis B vaccine at at day 1 and months 1 and 6.

Anti-HEV IgG and HBsAb were determined. Injection-site and systemic adverse events (AEs) were monitored for 30 days after any vaccination; serious AEs were monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people aged over 18 years old on the day of enrollment
* Negative in HBsAg,HBsAb and HBcAb.
* Judged as healthy and eligible for vaccination by the investigators through a selfreported medical history and some physical examinations.
* Able to understand this study information and willing to comply with all study requirements.
* Willing to participate in this study and sign informed consent form.

Exclusion Criteria:

* Pregnant or breastfeeding or planning on getting pregnant in the future 7 months
* Use of any investigational product or non-registered product (drug or vaccine)within 30 days preceding the first dose of the study vaccine or plan to use during the study period
* Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, exceptlocal treatment.
* Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine,or plan to use during the study period.
* Administration of any inactivated vaccines within 14 days preceding the first dose of the study or attenuated live vaccines within 21 days preceding the first dose of the study.
* Had a fever (axillary temperature over 38°C) within 3 days or acute illness requiring systemic antibiotics or antiviral treatment within 5 days before vaccination.
* Plan to participate in any other clinical trial during the study period
* Administration of HEV vaccine before the study.
* Immunodeficiency (such as HIV carriers), primary disease of important organs, malignant tumor,or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response).
* History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy,urticaria, dyspnea, angioneurotic edema or abdominal pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-08-25 (Actual)

PRIMARY OUTCOMES:
Adverse reactions/events | 7 months
  Measure solicited local adverse reactions within 7 days after each vaccination; Measure solicited systematic adverse reactions within 7 days after each vaccination; Measure unsolicited adverse reactions within 30 days after vaccination; Measure serious adverse events occurred throughout the study

SECONDARY OUTCOMES:
Immunogenicity | 7 months
  Measure anti-HEV antibody in serum samples at 7 month to evaluate the immunogenicity of the Hepatitis E vaccine. And measure the HBsAb in serum samples at 7 month to evaluate the immunogenicity of Hepatitis B vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Zhang, Principal Investigator — Beijing Chaoyang District CDC
Locations (1):
- Beijing Chaoyang District CDC, Beijing, Beijing Municipality, China